CLINICAL TRIAL: NCT05618366
Title: Phase I Trial of Tazemetostat in Combination With Venetoclax in Patients With Relapsed/Refractory Non-Hodgkin Lymphoma
Brief Title: Tazemetostat and Venetoclax in Relapsed/Refractory Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genentech, Inc. (Industry); Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-04024678
Record Dates: First submitted 2022-11-07; First posted 2022-11-16 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma, Non-Hodgkin; Diffuse Large B Cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — venetoclax; tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tazemetostat and Venetoclax (Experimental): All participants will receive a combination of oral 800 mg tazemetostat BID and oral venetoclax. Since this is a phase 1 trial, the dose of venetoclax will be determined by the investigators per a sequential dose escalation (3+3). Participants will be provided study drug in the form of pills to take at home. Study participants will need to regularly come to the clinic for blood work, imaging, and to monitor and side effects. Participants may receive study drug until their cancer progresses or for up to 24 months.
  Interventions: Drug: Venetoclax; Drug: Tazemetostat

INTERVENTIONS:
Drug: Venetoclax — Participants will receive oral venetoclax taken once per day. The dose will be between 200 and 800 mg daily, with the exact dose determined by the protocol.
  Other Names: Venclexta
Drug: Tazemetostat — Tazemetostat 800mg taken orally, twice daily.
  Other Names: Tazverik

SUMMARY:
The goal of this clinical trial is to learn about how a combination of tazemetostat and venetoclax in people with relapsed/refractory Non-Hodgkin Lymphoma (R/R NHL). The main questions that this trial aims to answer are what is the best dose of venetoclax to give with tazemetostat to people with R/R NHL; what types of side effects do people with R/R NHL get when taking venetoclax with tazemetostat; and what effects does this combination have on R/R NHL. Participants will need to take pills by mouth every day and regularly come to the clinic for blood work and imagining to monitor side effects and cancer progression. Participants may receive study drugs for up to 24 months.

DETAILED DESCRIPTION:
This a phase 1, single arm, non-randomized trial of tazemetostat in combination with venetoclax in participants with two types of relapsed/refractory non-Hodgkin lymphoma. The purpose of this study is to evaluate the safety of the combination of tazemetostat and venetoclax in patients with relapsed/refractory (R/R) Follicular Lymphoma (FL) and Diffuse Large B-cell Lymphoma (DLBCL).

This trial will be conducted in two parts. To evaluate the safety of the combination of tazemetostat and venetoclax in patients with relapsed/refractory (R/R) Follicular Lymphoma (FL) and Diffuse Large B-cell Lymphoma (DLBCL) we will conduct a phase I trial in two parts. In part one, we will perform a single-arm, open-label sequential dose escalation (3+3) of venetoclax in combination with tazemetostat, given at its recommended phase II dose (RP2D) of 800mg BID, to determine the maximum tolerated dose (MTD) of venetoclax. In part two, we will enroll two expansion cohorts (R/R DLBCL and R/R FL) to further characterize the safety and tolerability of the combination, and to estimate the preliminary efficacy.

Up to 18 participants will be enrolled in part 1 and 20 participants will be enrolled in part 2.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Adults aged ≥18
2. Require therapy as determined by the treating physician
3. Patients must have adequate organ and bone marrow function:

   * Absolute neutrophil count (ANC) ≥ 1 x 109/L without growth factor support (filgrastim or pegfilgrastim) for at least 14 days
   * Platelet count ≥75 x 109/L, evaluated at least 7 days after last platelet transfusion
   * Hemoglobin ≥9.0g/dL, independent of transfusion
   * Total bilirubin < 1.5 x's the upper limit of the normal range (ULN), except Gilbert's disease
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x's ULN.
   * Calculated creatinine clearance according to the Cockcroft-Gault equation. ≥ 40 mL/min
4. ECOG PS 0-2
5. Ability and willingness to provide signed Informed Consent Form
6. Ability and willingness to comply with the requirements of the study protocol
7. Measurable disease (defined as ≥ 1.5cm in diameter) In addition, patients must meet the following conditions for enrollment based on whether they have DLBCL or FL.

R/R DLBCL Cohort:

1. Histologically confirmed, biopsy-proven diagnosis of DLBCL (as determined by WHO standard classification criteria).

   Please note: Transformed DLBCL patients are eligible, with the exception of Richter's transformation.
2. Subjects must have received at least two prior lines of therapy for lymphoma with evidence of disease progression.
3. Subjects are eligible if they have progressed after ASCT OR if they are ineligible for ASCT, as determined by their treating physician.

R/R FL Cohort:

1. Histologically confirmed, biopsy-proven diagnosis of FL
2. Subjects are eligible if they have progressed after two or more lines of therapy for lymphoma or have no satisfactory treatment alternatives

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac ventricular arrhythmia.
2. Known hypersensitivity to any of the study drugs
3. History of other malignancy that could affect compliance with the protocol or interpretation of results

   a. Patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are generally eligible. Patients with a malignancy that has been treated, but not with curative intent, will also be excluded, unless the malignancy has been in remission without treatment for 2 years prior to enrollment.
4. Known CNS involvement at diagnosis (CNS evaluation not required in the absence of clinical suspicion)
5. Richter's transformation from CLL
6. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal).
7. Major surgery within 3 weeks prior to the start of study treatment
8. Venous thrombosis or pulmonary embolism within the last 3 months before starting study; whereas subjects greater than 3 months since deep vein thrombosis/pulmonary embolism are eligible but are recommended to receive prophylaxis.
9. Uncontrolled infection with human immunodeficiency virus (HIV) or human T-cell leukemia virus 1
10. Pregnant or lactating
11. Patients capable of becoming pregnant or getting someone else pregnant must be willing to use highly effective birth control as described in Section 4.4
12. Malabsorption syndrome or other condition that precludes enteral route of administration Patients who meet any of the following criteria will be excluded from study entry:
13. Inability to swallow tablets
14. Known allergy to both xanthine oxidase inhibitors and rasburicase
15. Clinically significant history of liver disease, including but not limited to viral or other hepatitis, current alcohol abuse, or cirrhosis Note: Subjects with positive HBV core antibody or surface antigen are eligible as long as they have an undetectable HBV DNA PCR and are willing to undergo monthly DNA testing, and receive concurrent antiviral therapy with entecavir, tenofovir, or lamivudine, and continued for a minimum of 6 months after completion of therapy.
16. Active hepatitis C (defined as a positive HCV viral load)
17. Chronic use of moderate or strong CYP3A4 modulators (inhibitor or inducer) or any other prohibited medications. A washout period of 5 half-lives or 14 days, whichever is longer, is required prior to venetoclax or tazemetostat dosing if a prohibited medication is discontinued.
18. Chronic use of a P-gp inhibitor, or a P-gp substrate with a narrow therapeutic index (see Section 7.8). A washout period of 5 half-lives or 14 days, whichever is longer is required prior to venetoclax or tazemetostat dosing if a prohibited medication is discontinued.
19. Prior exposure to either tazemetostat or venetoclax
20. Has a prior history of T-LBL/T-ALL
21. Subjects who have undergone a solid organ transplant
22. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the subject's participation in this study OR interfere with their ability to receive study treatment or complete the study.
23. Requires the use of warfarin (because of potential drug-drug interactions that may potentially increase the exposure of warfarin)
24. Vaccination with live vaccines within 28 days prior to treatment
25. Consumed grapefruit or grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) determination (Part 1) | Day 0 to 28
  In part 1 of this study, participants will be assigned a dose of venetoclax following a (3+3) dose escalation design and monitored for dose-limiting toxicities (DLTs) during the first treatment cycle. Based on observed DLTs observed in each dose level cohort, the maximum-tolerated dose will be determined. The # of patients experiencing a DLT among the evaluable patients for each dose level in part 1 will be tabulated.
Number of participants who experience dose-limiting toxicities (DLTs) | Day 0 to 28
  In part 1 of this study, participants will be assigned a dose of venetoclax following a (3+3) dose escalation design and monitored for dose-limiting toxicities (DLTs) during the first treatment cycle. Dose limiting toxicity (DLT) will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0).
Number of participants who experience adverse events (AEs), from baseline to 30 days after the last dose of study drug, as assessed by CTCAE v5.0 | Baseline through 25 months
  The safety analysis population will consist of all enrolled patients who receive at least one dose of study drug. AEs and SAEs will be tabulated by type, grade, and attribution for all patients overall and by treatment group. For each patient, and within each type of toxicity, the patient will be counted only once at the highest grade of that toxicity. Participants will be evaluated for AEs/SAEs from the time they sign the informed consent form until 30 days after their last dose of study drug.
Number of adverse events (AEs) by severity from baseline to 30 days, after the last dose of study drug as assessed, by CTCAE v5.0 | Baseline through 25 months
  The safety analysis population will consist of all enrolled patients who receive at least one dose of study drug. AEs and SAEs will be tabulated by type, grade, and attribution for all patients overall and by treatment group. For each patient, and within each type of toxicity, the patient will be counted only once at the highest grade of that toxicity. Participants will be evaluated for AEs/SAEs from the time they sign the informed consent form until 30 days after their last dose of study drug.

SECONDARY OUTCOMES:
Number of Participants who Achieve Complete Response (CR) | Day 0 through 24 months
  CR will be assessed for all evaluable patients in parts 1+2 according to Lugano response criteria.
Number of Participants who Achieve Partial Response (PR) | Day 0 through 24 months
  PR will be assessed for all evaluable patients in parts 1+2 according to Lugano response criteria.
Overall Response Rate (ORR) | Day 0 through 24 months
  The ORR response rate is the proportion of patients with a best overall response of either complete response (CR) or partial response (PR) among all evaluable patients. ORR, CR, and PR will be assessed for all evaluable patients in parts 1+2 according to Lugano response criteria. The best overall response is the best response recorded from the start of treatment until progressive disease.
Duration of Response (DoR) | From date of treatment initiation until the date of first documented progression or date of death from any cause, whichever came first, as assessed at 5 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or PD is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started).
  The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.
  Duration of stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started.
Progression-Free Survival | From date of treatment initiation until the date of first documented progression or date of death from any cause, whichever came first, as assessed at 5 years
  PFS is defined as the duration of time from start of treatment to time of documentation of progression or death from any cause.
Overall Survival (OS) | From date of treatment initiation until the date of death from any cause, as assessed at 5 years
  OS is defined as the duration of time from start of treatment to death from any cause.
Mean Change in Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Score from Baseline to End of Treatment | Baseline; at the start of Cycle 4 (a cycle is 28 days); at the start of Cycle 7; and End of Treatment (treatment will continue until disease progression or unacceptable toxicity for a maximum of approximately 2 years)
  FACT-Lym is a 42 item questionnaire that includes questions on physical well-being, social/family well-being, emotional well-being, functional well-being, and lymphoma symptoms over the past 7 days. Each response is measured on a 5 point Likert-type scale. Scores can range from 0 to 168 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Roth, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine/NewYork-Presberteryian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No